CLINICAL TRIAL: NCT02054832
Title: A Comparison of Quality of Sleep and Quality of Life in Patients With Glycogen Storage Disease on Standard and Modified Uncooked Cornstarch
Brief Title: Sleep and Quality of Life in Patients With Glycogen Storage Disease on Standard Versus Modified Uncooked Cornstarch
Status: Completed | Type: Observational
Sponsor: John Mitchell (Other)
Responsible Party: Sponsor-Investigator, John Mitchell, Division Head, Endocrinology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 12-337-PED
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Glycogen Storage Disease Type IA; Glycogen Storage Disease Type IB; Glycogen Storage Disease Type III; Glycogen Storage Disease Type 0
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease; Glycogen Storage Disease IB; Glycogen Storage Disease Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glycosade: A prospective cohort design will be used to assess the impact on sleep and continue to monitor safety of Glycosade.
  Interventions: Dietary Supplement: Glycosade

INTERVENTIONS:
Dietary Supplement: Glycosade

SUMMARY:
The aim of the present study is to determine if there is a change in quality and quantity of sleep perceived by adults and children with GSD and their parents while starting a modified UCCS (Glycosade) to prevent nocturnal hypoglycemia. The investigators also aim to evaluate if there is a change in quality of life perceived by adults and children and their parents with Glycosade.

DETAILED DESCRIPTION:
This is a prospective cohort study. Patients above 2 years old and their parents (for children only) will be enrolled during their usual follow-up. Parents will be asked to complete a quality of sleep questionnaire (as it pertains to both child and parent) relating to the past month on their current dietary regimen (standard UCCS) and a quality of life questionnaire (as it pertains to the child only). Parents will then complete a sleep diary (for both child and parent) and both child and parent will wear an actigraph that will record movements during sleep over a 1 week period. Adult GSD patients will complete their own questionnaires. Following this first assessment, they will be hospitalised over a 24 hour period as part of standard of care to start the modified UCCS, Glycosade, under supervision and with a continuous glucose monitoring (CGM) sensor. Following hospitalization, the family will return home. Glucose will be monitored with the aid of the CGM sensor for 5 to 7 days. The actigraphy and the sleep diary will be repeated after 2 weeks (for 1 week) while on Glycosade. One month after starting the modified UCCS, questionnaires on quality of sleep and quality of life will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ≥ 2 years old with a diagnostic of GSD 0, I, III, VI, IX or XI based on a liver biopsy, mutation in the appropriate gene or clinical evidence of GSD with a positive familial history
* Medical history of fasting hypoglycemia
* Currently taking standard UCCS
* With a stable condition
* Followed in GSD clinics at the Montreal Children's Hospital and the Hôpital St-Luc
* With informed consent obtained

Exclusion Criteria:

* Continuous overnight feeds

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Glycogen Storage Disease taking uncooked cornstarch to prevent hypoglycemia followed at the Montreal Children's Hospital and St-Luc Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The aim of the present study is to determine if there is a change in quality and quantity of sleep perceived by GSD adults and children and their parents while starting a modified UCCS (Glycosade) to prevent nocturnal hypoglycaemia. | 2 weeks
  Parents will be asked to complete a quality of sleep questionnaire (as it pertains to both child and parent) relating to the past month on their current dietary regimen (standard UCCS). Parents will also complete a sleep diary (for both child and parent) and both child and parent will wear an actigraph that will record movements during sleep over a 1 week period prior to Glycosade. The actigraphy and the sleep diary will be repeated after 2 weeks (for 2 weeks) while on Glycosade. The quality of sleep questionnaire will be repeated after 1 month on Glycosade. Adult GSD patients will complete their own questionnaires.

SECONDARY OUTCOMES:
To evaluate if there is a change in quality of life perceived by GSD adults and children and their parents with Glycosade. | 1 month
  Parents (as it pertains to their child) and adult patients will be asked to complete quality of life questionnaire prior to Glycosade and 1 month after starting this new diet.

OTHER OUTCOMES:
To describe the variability in glucose fluctuations with Glycosade using a CGM sensor. | 1 week
  Glucose will be monitored with the aid of the CGM sensor for 5 to 7 days while starting Glycosade.
To establish if metabolic control is maintained using Glycosade. | 24 hours
  Metabolic control in hospital after starting Glycosade will be defined as the absence of deterioration of biochemical data at the end of fast compared to during the fast.
To evaluate the safety profile of Glycosade, based on the frequency of side effects, e.g. gastrointestinal side effects while receiving Glycosade. | 1 month
  Subjects will be constantly monitored for adverse events throughout the study. They will be asked to keep a diary to document side effects while receiving Glycosade. They will also be asked at each visit whether they experienced any known or unknown side effects.
To assess the acceptability/palatability of Glycosade. | 1 month
  Patient report (or parent report on behalf of child) of palatability at 4 weeks after starting Glycosade compared to their previous regimen.

CONTACTS AND LOCATIONS:
Overall Officials: John J Mitchell, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- Montreal Children's hospital, Montreal, Quebec, Canada